CLINICAL TRIAL: NCT07402460
Title: Effects of a Programmed Reflexology Therapy on Sleep Quality, Insomnia, and Fatigue Among Individuals With Poor Sleep Quality: Evidence for Autonomic Nervous System Modulation
Brief Title: Effects of a Programmed Reflexology Therapy on Sleep Quality, Insomnia, Fatigue, and Heart Rate Variability Among Individuals With Poor Sleep Quality
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Wen Ching Huang, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C113172
Record Dates: First submitted 2026-01-14; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Poor Sleep Quality
Keywords: Poor sleep quality; Pittsburgh Sleep Quality Index; Foot reflexology; Heart rate variability; Autonomic nervous system

STUDY DESIGN:
Intervention Model Description: This study employs a randomized crossover interventional study model. All participants receive both interventions-manual reflexology treatment and mechanical foot massage-administered in two separate intervention periods. The order of interventions is randomized to minimize order and carryover effects, allowing each participant to serve as their own control. Each intervention period lasts six weeks and is separated by a washout interval to reduce potential residual effects from the preceding intervention. This design enhances internal validity and enables direct comparison of the effects of the two interventions on sleep-related outcomes and autonomic nervous system function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual reflexology treatment (Experimental): Participants assigned to the manual reflexology treatment arm receive a structured, therapist-delivered foot reflexology intervention administered once weekly for 6 weeks. Each session lasts approximately 30-40 minutes and follows a standardized protocol based on predefined reflex zones of both feet. The intervention includes systematic relaxation techniques, stimulation of whole-foot reflex areas, and targeted reinforcement of reflex zones associated with sleep regulation and autonomic nervous system function. All treatments are delivered by a certified reflexology practitioner in a quiet, controlled environment, with procedures standardized according to the Template for Intervention Description and Replication (TIDieR) framework to ensure consistency and reproducibility.
  Interventions: Behavioral: manual reflexology treatment; Behavioral: Feet massage using an electric massager (FEM)
- mechanical foot massage (Active Comparator): The participants received feet massage using an electric massager (Model HY-703, HUEI YEH, Taipei, Taiwan). Each session lasted 30 minutes and was conducted using the device's pre-set "fatigue relief" mode, which applied medium-intensity pressure combined with a mild heating function. The massage covered the following regions with different mechanical actions. (1) Plantar region (sole of the foot): Targeted zones included the thoracic, abdominal, and pelvic areas. The massage's methods were delivered using rolling, pressing, squeezing, and vibration techniques. (2) Medial and lateral sides of the foot: These areas were stimulated through squeezing, pressing, and vibration. (3) Dorsal foot region (top of the foot): This region was massaged using squeezing, pressing, and vibration. (4) Calf region: The device provided massage through squeezing, pressing, and vibration to promote circulation and muscle relaxation.
  Interventions: Behavioral: manual reflexology treatment; Behavioral: Feet massage using an electric massager (FEM)

INTERVENTIONS:
Behavioral: manual reflexology treatment — The manual reflexology procedure was carried out following a standardized sequence, targeting specific foot reflex zones. The detailed steps were as follows:
  1. Preparation: All participants were positioned in a semi-recumbent supine posture on a treatment bed, with appropriate towel draping to ensure comfort and privacy. The massage bed and chair were disinfected with 75% alcohol and covered with a clean foot towel.
  2. Foot Relaxation Techniques: The treatment began with relaxation techniques (e.g., friction and oscillation) applied first to the left foot, followed by the right.
  3. Reflex Zone Stimulation Techniques: Five core massage techniques-pressing, kneading, pushing, scraping, and acupressure-were applied systematically across different reflex zones, as described below:
  I. Toe Region (2 min/foot): Brain, frontal lobe, pituitary gland, temples, cerebellum, nose, cervical area, eyes, ears, upper/lower jaw, tonsils, vocal cords, esophagus, and trachea.
  II. Medial Foot (2 min/
Behavioral: Feet massage using an electric massager (FEM) — Each session lasted 30 minutes and was conducted using the device's pre-set "fatigue relief" mode, which applied medium-intensity pressure combined with a mild heating function. The massage covered the following regions with different mechanical actions. (1) Plantar region (sole of the foot): Targeted zones included the thoracic, abdominal, and pelvic areas. The massage's methods were delivered using rolling, pressing, squeezing, and vibration techniques. (2) Medial and lateral sides of the foot: These areas were stimulated through squeezing, pressing, and vibration. (3) Dorsal foot region (top of the foot): This region was massaged using squeezing, pressing, and vibration. (4) Calf region: The device provided massage through squeezing, pressing, and vibration to promote circulation and muscle relaxation. All participants received the same standardized massage setting to ensure consistency throughout the intervention period.

SUMMARY:
The goal of this clinical trial is to evaluate whether a structured reflexology therapy can improve sleep, reduce insomnia severity, and alleviate fatigue in adults with poor sleep quality, and to understand how it affects autonomic nervous system function. The main questions it aims to answer are:

* Can manual reflexology treatment improve sleep quality as measured by standardized sleep assessments?
* Can manual reflexology influence physiological measures of autonomic function (such as heart rate and heart rate variability)?

Researchers will compare the effects of a manual reflexology intervention to those of a mechanical foot massage to determine which approach is more effective in improving sleep, reducing insomnia severity, and enhancing fatigue and autonomic balance.

Participants will be asked to:

* Undergo weekly sessions of manual reflexology therapy for six weeks, and
* Undergo weekly sessions using mechanical foot massage equipment for six weeks, with heart rate, heart rate variability, and sleep and fatigue questionnaires measured before and after each intervention period.

DETAILED DESCRIPTION:
Poor sleep quality is a common health concern associated with impaired autonomic nervous system regulation and increased risk of physical and psychological disorders. Complementary therapies, such as foot reflexology, are widely used to promote relaxation and improve sleep; however, evidence regarding their physiological effects and comparative effectiveness remains limited. This study was designed to examine whether a structured manual reflexology treatment can improve sleep-related outcomes and autonomic nervous system function in adults with poor sleep quality, compared with mechanical foot massage.

Participants enrolled in this study undergo two different foot-based interventions-manual reflexology treatment and mechanical foot massage-delivered in separate intervention periods. Each intervention period lasts six weeks, with one session per week. The order of interventions is assigned using a randomized crossover design, allowing each participant to receive both treatments while minimizing individual differences.

Manual reflexology sessions are delivered by a trained practitioner following a standardized and reproducible protocol, which targets specific foot reflex zones associated with relaxation and autonomic regulation. Mechanical foot massage sessions are conducted using commercially available foot massage equipment under standardized conditions. Both interventions are designed to be non-invasive and well tolerated.

Throughout the study, participants' physiological responses are monitored using non-invasive measures of heart rate and heart rate variability, which provide insight into autonomic nervous system activity. In addition, participants complete validated questionnaires assessing sleep quality, insomnia severity, and fatigue. By comparing changes observed after each intervention, this study aims to clarify whether manual reflexology offers added benefits over mechanical massage and to explore the potential role of autonomic modulation in improving sleep-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. . Aged between 40 and 80 years.
2. . Had no prior experience with, or had not regularly received, feet massage treatments.
3. . Had a global score greater than 10 on the PSQI, indicating poor sleep quality.

Exclusion Criteria:

1. . Presence of bacterial or viral infections on the feet.
2. . Acute infectious diseases, bleeding or coagulation disorders, psychiatric conditions, open wounds, or bone fractures.
3. . Conditions such as extreme fatigue, physical weakness, alcohol intoxication, or long-term bedridden status that prevented attendance at the study site.
4. . Lower limb amputation or significant limb deficiency.
5. . Employment involving rotating or shift work.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | Baseline and after 6 weeks of each intervention period
  Sleep quality is assessed using the Pittsburgh Sleep Quality Index (PSQI), a validated self-reported questionnaire that evaluates overall sleep quality and seven component domains, including sleep latency, duration, efficiency, disturbances, use of sleep medication, and daytime dysfunction. Higher scores indicate poorer sleep quality.

SECONDARY OUTCOMES:
Insomnia Severity | Baseline and after 6 weeks of each intervention period
  Insomnia severity is measured using the Insomnia Severity Index (ISI), a validated 7-item self-report questionnaire assessing perceived severity of insomnia symptoms, sleep satisfaction, daytime impairment, and distress related to sleep difficulties. Total scores range from 0 to 28, with higher scores indicating greater insomnia severity.
Fatigue Severity | Baseline and after 6 weeks of each intervention period
  Fatigue is assessed using the Fatigue Assessment Scale (FAS), a validated self-reported questionnaire evaluating both physical and mental fatigue. Higher total scores indicate greater perceived fatigue.
Autonomic Nervous System Function (Heart Rate Variability) | Baseline and immediately after intervention at week 1 and week 6 of each intervention period
  Autonomic nervous system function is evaluated using heart rate variability (HRV) derived from electrocardiogram recordings. Time-domain indices (SDNN, RMSSD, pNN50) and frequency-domain indices (LF, HF, LF/HF ratio) are analyzed to reflect sympathetic and parasympathetic modulation. Higher RMSSD, pNN50, and HF values indicate greater parasympathetic activity.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cai DC, Chen CY, Lo TY. Foot Reflexology: Recent Research Trends and Prospects. Healthcare (Basel). 2022 Dec 20;11(1):9. doi: 10.3390/healthcare11010009. PMID 36611469

DOCUMENTS (1):
  • Statistical Analysis Plan: Cover page-Statistical Analysis Plan (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT07402460/SAP_000.pdf